CLINICAL TRIAL: NCT06544408
Title: Rapid Treatment of PTSD With Accelerated Non-Invasive Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, F. Andrew Kozel, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00005179; CDMRP-TP230396 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder; Traumatic Brain Injury
Keywords: PTSD; TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding Procedures The participants, PI, Research Staff involved in TMS treatment, and staff performing the study procedures will be blinded to the participant's dl-PFC protocol assignment throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Arm 1: active left dl-PFC accel-TMS (Active Comparator): Acute Phase: Eligible participants will be randomized into one of the three treatment groups: active left dl-PFC accel-TMS vs. active dm-PFC accel-TMS vs. sham dl-PFC/dm-PFC accel TMS
  Interventions: Device: Cool B70 AP Coil - Active (dl-PFC)
- Arm 2:active dm-PFC accel-TMS (Active Comparator): Acute Phase: Eligible participants will be randomized into one of the three treatment groups: active left dl-PFC accel-TMS vs. active dm-PFC accel-TMS vs. sham dl-PFC/dm-PFC accel TMS
  Interventions: Device: Cool D-B80 AP Coil - Active (dm-PFC)
- Arm 3 - sham accel-TMS dl-PFC (Sham Comparator): Acute Phase: Eligible participants will be randomized into one of the three treatment groups: active left dl-PFC accel-TMS vs. active dm-PFC accel-TMS vs. sham dl-PFC/dm-PFC accel TMS
  Interventions: Device: Cool B70 AP Coil- Sham (dl-PFC)
- Arm 4: sham accel -TMS dm-PFC (Sham Comparator): Acute Phase: Eligible participants will be randomized into one of the three treatment groups: active left dl-PFC accel-TMS vs. active dm-PFC accel-TMS vs. sham dl-PFC/dm-PFC accel TMS
  Interventions: Device: Cool D-B80 AP Coil - Sham (dm-PFC)
- Arm 5 (Active Comparator): Extension phase, all participants will receive active left dl-PFC accel-TMS.
  Interventions: Device: Cool B70 Treatment Coil - Active Only

INTERVENTIONS:
Device: Cool B70 AP Coil - Active (dl-PFC) — One side of the coil is the active and the other is sham. The B70 AP coil will be positioned over the left dorsolateral prefrontal cortex (dl-PFC).
  Arms: Arm 1: active left dl-PFC accel-TMS
Device: Cool B70 AP Coil- Sham (dl-PFC) — One side of the coil is the active and the other is sham. The B70 AP coil will be positioned over the left dorsolateral prefrontal cortex (dl-PFC).
  Arms: Arm 3 - sham accel-TMS dl-PFC
Device: Cool D-B80 AP Coil - Active (dm-PFC) — One side of the coil is the active and the other is sham. The cool D-B80 AP coil will be positioned over the midline (bilateral) dorsal medial prefrontal cortex (dmPFC) using location 25.8% distance from nasion to inion.
  Arms: Arm 2:active dm-PFC accel-TMS
Device: Cool D-B80 AP Coil - Sham (dm-PFC) — One side of the coil is the active and the other is sham. The cool D-B80 AP coil will be positioned over the midline (bilateral) dorsal medial prefrontal cortex (dmPFC) using location 25.8% distance from nasion to inion.
  Arms: Arm 4: sham accel -TMS dm-PFC
Device: Cool B70 Treatment Coil - Active Only — The treatment will be the same as the left dl-PFC accel-TMS dl-PFC except that the Cool B70 Treatment coil only has an active treatment coil.
  Arms: Arm 5

SUMMARY:
This study will test the clinical efficacy of an accelerated TMS (accel-TMS) protocol that rapidly addresses PTSD symptoms with 1 week (25 sessions over 5 days) of condensed treatment.

DETAILED DESCRIPTION:
This study will have three phases: an acute phase (1 week of treatments), an extension phase (second week of treatments), and a long-term observational follow-up phase of 6 months.

The acute phase will be a three-arm randomized sham-controlled trial with: Arm 1 = active left dl-PFC accel-TMS; Arm 2 = active dm-PFC accel-TMS; and Arm 3 = sham accel-TMS (half with sham dl-PFC and half with sham dm-PFC coil positioning).

In the subsequent extension phase, all participants will receive active left dl-PFC accel-TMS. For the follow-up phase, clinical outcomes will be assessed at 1-month, 3-months, and 6-months. The primary outcome measure will be the CAPS-5.

A range of other secondary outcome measures will also be included.

ELIGIBILITY:
Inclusion:

1. Adults age 18 years to 65 years old.
2. Meets DSM-5 criteria for PTSD with a PCL-5 score > 33
3. No changes in psychotropic medication (if taking psychotropic medication) and/or changes in supportive psychotherapy for 1 month prior to initial visit; and clinically appropriate to maintain stable treatment regimen for duration of trial.
4. Clinically competent to give informed written consent and ability to understand study procedures and to comply with them for the entire length of the study

Exclusion:

1. Medical contraindication for neuromodulation (e.g., ferrous metal in head, seizure disorder, brain tumor, stroke, aneurysm, multiple sclerosis, etc.).
2. Active substance use disorder in last 3 months or any current substance use that puts the participant at increased risk or significant impairment.
3. Dementia or other cognitive disorder making unable to engage in treatment.
4. Any history or diagnosis of Schizophrenia, Schizoaffective Disorder, Delusional Disorder or other psychotic illness that precludes safe participation in trial.
5. Suicidal risk that precludes safe participation defined as clinical impression that the participant is at significant risk for suicide.
6. OCD cannot be the primary disorder but can have OCD symptoms.
7. Inability to stop taking any medication that significantly lowers the seizure threshold (e.g., tricyclic antidepressants, clozapine, etc.)
8. Current, planned, or suspected pregnancy
9. Unstable medical conditions or any current medical condition that could preclude being able to safely participate in TMS treatment (e.g., unstable metabolic abnormality, unstable angina, etc.)
10. Severe Traumatic Brain Injury
11. We will exclude non-English speakers because of the need for rapid communication during the delivery of treatments.
12. Significant ongoing litigation or claims that impact research activities, as determined by the research study team. (Research may especially be impacted when mental health or pain is being evaluated for litigation or claims, such as civil and criminal cases, disability claims and worker's compensation).
13. Prior known active TMS of dorsolateral prefrontal cortex or dorsomedial prefrontal cortex or electroconvulsive therapy (ECT) -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) to determine left dl-PFC accel-TMS efficacy | Assessment of symptoms during the preceding week.
  CAPS-V is a 30-item clinical interview used to diagnose PTSD as well as monitor PTSD symptoms. Questions address the traumatic event(s), symptom duration, subjective distress, impact on functioning, dissociation, and symptom improvement since last evaluation.
  During the Acute Phase, CAPS-V will be used to determine the rapid efficacy of left dl-PFC accel-TMS compared to sham accel-TMS at approximately one-week post-treatment.
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) to determine dm-PFC accel-TMS efficacy | Assessment of symptoms during the preceding week.
  A 30-item clinical interview used to diagnose PTSD as well as monitor PTSD symptoms. Questions address the traumatic event(s), symptom duration, subjective distress, impact on functioning, dissociation, and symptom improvement since last evaluation.
  During the Acute Phase, CAPS-V will be used to determine the rapid efficacy of dm-PFC accel-TMS compared to sham accel-TMS at approximately one-week post-treatment
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) to determine superior symptom reduction | Assessment of symptoms during the preceding week.
  A 30-item clinical interview used to diagnose PTSD as well as monitor PTSD symptoms. Questions address the traumatic event(s), symptom duration, subjective distress, impact on functioning, dissociation, and symptom improvement since last evaluation.
  During the Extension Phase, CAPS-V will be used to determine whether an additional week of left dl-PFC accel-TMS provides superior reduction of PTSD symptoms compared to one week of left dl-PFC accel-TMS.

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) to characterize durability of accel-TMS effects | Assessment of symptoms during the preceding week before each follow-up visit.
  A 30-item clinical interview used to diagnose PTSD as well as monitor PTSD symptoms. Questions address the traumatic event(s), symptom duration, subjective distress, impact on functioning, dissociation, and symptom improvement since last evaluation.
  During Follow-Up Phase to characterize the durability of accel-TMS effects on PTSD symptoms at 1-month, 3-months, and 6-months post treatment.
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) to determine superior outcomes between active left dl-PFC and active dm-PFC accel-TMS | Assessment of symptoms during the preceding week.
  A 30-item clinical interview used to diagnose PTSD as well as monitor PTSD symptoms. Questions address the traumatic event(s), symptom duration, subjective distress, impact on functioning, dissociation, and symptom improvement since last evaluation.
  During the Acute Phase to determine whether active left dl-PFC or active dm-PFC accel-TMS produces superior outcomes for PTSD symptoms
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) to determine added benefit during Extension | Assessment of symptoms during the preceding week.
  A 30-item clinical interview used to diagnose PTSD as well as monitor PTSD symptoms. Questions address the traumatic event(s), symptom duration, subjective distress, impact on functioning, dissociation, and symptom improvement since last evaluation.
  During the Extension Phase to determine whether an additional week of open left dl-PFC accel-TMS will provide added benefit to those participants that received active dm-PFC accel-TMS (i.e., targeting 2 brain regions versus 1 brain region).

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Kozel, MD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT06544408/ICF_001.pdf